CLINICAL TRIAL: NCT01799161
Title: Phase 1 Study of the Combination of gp96-Ig Cell Based Lung Cancer Vaccine With Suppression of Adenosinergic Pathways With Theophylline and Oxygen for the Treatment of Non-Small Cell Lung Cancer (NSCLC) Patients With Advanced (Stage IIIB), Relapsed or Metastatic (Stage IV) Disease Who Have Failed Palliative Therapy.
Brief Title: Combination of gp96-Ig Vaccine, Theophylline and Oxygen for the Treatment of Patients With Advanced, Relapsed or Metastatic Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Eckhard Podack (Other)
Responsible Party: Sponsor-Investigator, Eckhard Podack, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20110847
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Non-Small Cell Lung Cancer; Non-small-cell Lung Carcinoma; Lung Cancer; NSCLC
Keywords: NSCLC; Lung Cancer; gp96; gp96 Vaccine; AD100-gp96Ig-HLA A1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — glucose-regulated proteins; Theophylline; Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DS-1 (Active Comparator): 6 week course of gp96 Vaccine: >= 4 x 10^7 cells twice monthly on Day 1. Up to 3 courses, 9 vaccinations.
  Interventions: Biological: gp96-Ig Vaccine; Drug: Theophylline; Other: Oxygen; Procedure: Immunologic Evaluation
- DS-2 (Active Comparator): 6 week course of gp96 Vaccine: >= 2 x 10^7 cells weekly on Day 1. Up to 3 courses, 18 vaccinations.
  Interventions: Biological: gp96-Ig Vaccine; Drug: Theophylline; Other: Oxygen; Procedure: Immunologic Evaluation
- DS-3 (Active Comparator): 6 week course of gp96 Vaccine: >= 1 x 10^7 cells twice weekly on Days 1 and 4. Up to 3 courses, 36 vaccinations.
  Interventions: Biological: gp96-Ig Vaccine; Drug: Theophylline; Other: Oxygen; Procedure: Immunologic Evaluation

INTERVENTIONS:
Biological: gp96-Ig Vaccine
  Other Names: gp96; AD100-A1-gp96Ig vaccine; Short gp96 Vaccine; gp96IG and HLA A1 Transfected NSCLC Cell Line
Drug: Theophylline — 300 mg capsule daily of Theophylline during 1st course, then adjusted dose
  Other Names: dimethylxanthine
Other: Oxygen — 24-hr oxygen delivered via nasal cannula or oxygen mask during 1st course, then adjusted dose.
  Other Names: O2
Procedure: Immunologic Evaluation — Frequency of IFN-y,CD8 cells in response to vaccine in available tumor samples Blood draw to assess immunological response [frequency of CD4+, FoxP3 (Treg), et al] in treated patients.
  Other Names: Peripheral Blood Sample; Tumor Sample

SUMMARY:
NSCLC tumors are appropriate targets for active immunotherapy, because they are non-immunogenic, which indicates that NSCLC does not stimulate a spontaneous immune response.

NSCLC tumor-secreted gp96-Ig is an ideal vaccine because it combines adjuvant activity with polyvalent peptide specificity. Tumor secreted gp96 activates dendritic cells (DC), natural killer cells (NK) and cytotoxic T lymphocytes (CTL). Tumor cells can be killed by NK-specific mechanisms, by promiscuous killing of CD8 CTL through NKG2D, and by MHC restricted CD8 CTL activity. The activation of DC and NK by tumor secreted gp96 may also counteract the generation of immuno-suppressive CD4 regulatory cells.

Suppression of adenosinergic pathways by oxygen and theophylline in combination with immunotherapy will improve tumor rejection.

Allogeneic, gp96-Ig secreting tumor cells used as vaccine are expected to generate NK and CTL with activity to the patient's autologous tumor.

DETAILED DESCRIPTION:
This is a proof of principle trial investigating a heat shock protein gp96 Ig-secreting, allogeneic tumor cell-vaccine (gp96-Ig vaccine) administered in combination with suppression of adenosinergic pathways by oxygen and Theophylline to patients with non-small cell lung cancer (NSCLC). Allogeneic, cultured lung adenocarcinoma cells transfected with HLA A1 and gp96-Ig will be irradiated and injected intradermally into patients suffering from advanced, relapsed, or metastatic NSCLC. HLA matching is not required. Safety and immunogenicity of the combined treatment will be studied in three patient cohorts that will receive twice monthly, weekly or twice weekly vaccination plus Theophylline and oxygen.

Immune response to vaccination of patients will be measured by determining adenocarcinoma-specific CD8 CTL precursor frequencies. ELI-spot assay for interferon-y (IFN-y) will be done to measure cytotoxic function of CD8 cells challenged in vitro with vaccine cells or autologous tumor cells. Multiparameter flow cytometry of CD8 and CD4 cells will be carried out to assess functional characteristics and to assess adenosine receptor levels and expression of hypoxia inducible factor-1alpha.

Patients will be randomized in equal allocation (1:1:1) to one of three dose-schedule (DS) cohorts defined by the frequency of vaccination. All patients will receive a total course dose of gp96 vaccine. A total of 36 patients, 12 per DS cohort, will be enrolled. We expect to accrue at a rate of two patients per month except at the onset of study when successive enrollment will be spaced to allow observation of first course toxicity in the first several patients. (See Section 3.3.4 for details.) Patients will be followed for a minimum of one year, thus study duration is expected to be three years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC (squamous, adeno-, large cell anaplastic, bronchoalveolar, and non-small cell carcinoma NOS): stage IIIB with malignant pleural effusion, stage IV, or recurrent disease.
* At least one site of measurable disease.
* Brain metastasis if present and treated must be stable by CT scan or MRI for at least 4 weeks after treatment.
* Patient must have received and failed at least one line of palliative therapy (chemotherapy or biological therapy)
* Age >= 18 years.
* ECOG performance status 0-2.
* Life expectancy >= 3 months.
* Laboratory parameters

  * Hemoglobin levels >= 10.0 (transfusions allowed if necessary).
  * ANC >= 1,500.
  * Platelets >= 100k.
  * Creatinine clearance >= 50 ml/min.
  * Total and direct bilirubin: < 3.0 x upper institution limit for normal.
  * Liver function tests: AST, ALT, and AlkP < 3.0 x upper institution limit for normal.
  * Signed informed consent.

Exclusion Criteria:

* Active or symptomatic cardiac disease such as congestive heart failure, angina pectoris or recent myocardial infarction. Patients with history of these conditions who are stable taking cardiac medications will also be excluded.
* Pregnant or lactating women (negative test for pregnancy is required of women of childbearing potential).
* Known HIV infection.
* Uncontrolled or untreated brain or spinal cord metastases.
* Active infection.
* Concomitant steroid or other immunosuppressive therapy.
* Other active malignancies present within the past three years, except for basal and/or squamous cell carcinoma(s) or in situ cervical cancer.
* Meningeal carcinomatosis.
* Chemotherapy, radiation therapy, or other anti-tumor therapy during the last three weeks.
* Immune deficiency syndromes, including the following: rheumatoid arthritis, systemic lupus erythematousus, Sjogren's disease, sarcoidosis, vasculitis, polymyositis, glomerulonephritis.
* Compromised lung function:

  * FeV1 < 30% of the predicted value, or
  * DLCO < 30% of the predicted value, or
  * PCO2 > 45 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events Experienced by Patients Receiving Study Treatment | 36 months
  Evaluation of the safety of administering a heat shock protein gp96-Ig-secreting allogeneic tumor cell-vaccine (gp96-Ig vaccine) in combination with oxygen and theophylline in patients with advanced NSCLC.

SECONDARY OUTCOMES:
Immune response to vaccination | 36 months
Clinical Response to gp96-Ig Vaccination | 36 months
  Clinical Response to gp96-Ig Vaccination measured by CT scan and RECIST criteria v 1.1.
Recommended Dose-schedule Combination for further testing | 36 Months
  The recommended Dose-schedule combination of gp96-Ig vaccine, Theophylline and Oxygen for NSCLC in further testing

CONTACTS AND LOCATIONS:
Overall Officials: Ikechukwu Akunyili, MD, Principal Investigator — University of Miami